CLINICAL TRIAL: NCT05953389
Title: An Exploratory, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Effect and Safety of Pitolisant in Children and Adolescents With Autism Spectrum Disorders
Brief Title: Proof of Concept Study on Pitolisant Effect on Autism Spectrum Disorders in Children and Adolescents
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P21-01 / BF2.649
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pitolisant (Experimental): One tablet of pitolisant 5 mg, two tablets of pitolisant 5 mg, one tablet of pitolisant 20 mg or two tablets of pitolisant 20 mg per day for 12 weeks.
  Interventions: Drug: Pitolisant
- Placebo (Placebo Comparator): One or two tablets of matching placebo per day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitolisant — histamine H3 receptor antagonist/inverse agonist
  Other Names: BF2.649
  Arms: Pitolisant
Drug: Placebo — Matching placebo of pitolisant tablets
  Arms: Placebo

SUMMARY:
Proof of concept, multicenter, randomized, double-blind, placebo-controlled, parallel-group, study to investigate the effect, safety, tolerability and pharmacokinetics of pitolisant in male children and adolescents with Autism Spectrum Disorders.

DETAILED DESCRIPTION:
First clinical study to assess the effect of BF2.649 in male children and adolescent with a diagnosis of Autism spectrum disorders according to DSM-5 criteria and confirmed by the Autism Diagnostic Observation Schedule (ADOS-2) or Autism Diagnostic Interview-Revised (ADI-R) over a 12-weeks period.

ELIGIBILITY:
Inclusion Criteria:

* Participants and their parent(s)/legal guardian(s) are willing and able to give informed assent and consent for participation in the study.
* Male children and adolescents aged from 6 to 17 inclusive for the duration of study participation.
* Diagnosis of autism spectrum disorders (ASD) as per the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria confirmed by the Autism Diagnostic Observation Schedule (ADOS-2) or the Autism Diagnostic Interview-Revised (ADI-R).
* Intelligence Quotient (IQ) ≥ 70 using Wechsler Intelligence Scale.
* Social Responsiveness Scale Second Edition (SRS-2) total T-score ≥ 66 at screening and baseline.

Exclusion Criteria:

* Previous genetic diagnosis of ASD-known "syndromic" ASD (e.g., Fragile X syndrome, Angelman syndrome, Prader-Willi, Rett's syndrome, tuberous sclerosis, Dup15q syndrome).
* History of suicidal behavior or suicidal ideation in the past 12 months, or a positive answer to questions 4 or 5 on the Columbia-Suicide-Severity Rating Scale (C-SSRS) at screening and/or baseline, and/or is a significant risk for suicidal behavior per investigator judgement.
* History or current diagnosis of epilepsy or any seizure occurring after the age of 5.
* Clinically significant deviation from normal on 12-lead ECG that results in an active medical problem, per investigator judgement or, with a corrected QT interval by Fridericia (QTcF) > 450ms at screening.
* Severe hepatic impairment (Child Pugh C) or with any other hepatic significant abnormality in the physical examination or alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) ≥ 2x Upper Limit of Normal (ULN) for age at laboratory results.

Ages: 6 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale Second Edition (SRS-2) total score | 12 weeks
  65-item informant-based rating scale designed specifically for use in Autism Spectrum Disorders to quantitatively measure an individual's ability to engage in emotionally appropriate reciprocal social behavior with higher scores indicating greater impairment.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale III (VABS III) total score | 12 weeks
  Instrument that measures socialization, communication, daily living skills, motor skills and maladaptive behavior of individuals with intellectual disabilities;
Incidence of Treatment-Emergent adverse events (AEs) as assessed by AEs collection | 12 weeks
  Safety assessment of pitolisant based on adverse events (AEs) reporting during the treatment pe

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bonnot, MD, Prof., Principal Investigator — Etablissement Public de Santé Barthélemy Durand, Sainte-Geneviève-des-Bois, France
Locations (15):
- France (3):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Nantes University Hospital, Nantes
  - CH le Rouvray, Sotteville-lès-Rouen
- Italy (9):
  - IRCCS-Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Istituto Scientifico IRCCS E. Medea, Bosisio Parini
  - Clinica Di Neuropsichiatria Infantile, Cagliari
  - IRCCS Fondazione Stella Maris, Calambrone
  - A.O.U Ospedali Riuniti di Foggia- Cardiologia (U.O.C), Foggia
  - IRCCS Centro Neurolesi Bonino Pulejo, Messina
  - Universita degli Studi di Napoli Federico II, Napoli
  - IRCCS Instituto Neurologico Casimiro Mondino, Pavia
  - Azienda ospedaliero-universitaria Senese, Siena
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
- Cognition Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No